CLINICAL TRIAL: NCT05778227
Title: Comparing the Dentin Conditioning Effect of Different Single and Combination Chelating Agents on Sealer Penetration and Dentin Erosion
Brief Title: Comparing Different Single and Combination Chelating Agents on Sealer Penetration and Dentin Erosion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sehrish Zubair, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: szubair
Record Dates: First submitted 2023-01-22; First posted 2023-03-21 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Root Canal Infection; Periapical Abscess; Irreversible Pulpitis; Apical Periodontitis
MeSH Terms: conditions — Periapical Abscess; Periapical Periodontitis | interventions — Edetic Acid; Etidronic Acid; Sodium Hypochlorite; maleic acid

STUDY DESIGN:
Intervention Model Description: Four group assigned with interventions and one control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study the participants are coded and the outcome assessor is blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Ethylene Diamine Tetra Acetic acid (Active Comparator): Final irrigation will be done with 5ml of EDTA for 1min which is the gold standard and compare it with experimental irrigants.
  Interventions: Drug: Ethylene Diamine Tetra Acetic acid
- smearOFF (Experimental): Final irrigation will be done with 5ml of EDTA for 1min which is the gold standard and compare it with experimental irrigants.
  Interventions: Drug: smearOFF
- Etidronic acid/ Sodium Hypochlorite (HEBP/NaOCl) (Experimental): During whole procedure of cleaning and shaping combination product of HEBP/NaOCl will be used
  Interventions: Drug: Etidronic acid /sodium hypochlorite
- Maleic acid (MA) (Experimental): Final irrigation of root canal treatment procedure will be done with 5ml of maleic acid for 1min.
  Interventions: Drug: Maleic acid
- Control group (No Intervention): Final irrigation of root canal treatment will be done with 0.9% saline.

INTERVENTIONS:
Drug: Ethylene Diamine Tetra Acetic acid — Final irrigation will be done with 5ml of EDTA for 1min which is the gold standard and compare it with experimental irrigants.
  Other Names: EDTA
  Arms: Ethylene Diamine Tetra Acetic acid
Drug: smearOFF — Final irrigation of root canal treatment procedure will be done with 5ml of smearOFF for 1min.
  Other Names: SOFF
  Arms: smearOFF
Drug: Etidronic acid /sodium hypochlorite — During whole procedure of cleaning and shaping combination product of HEBP/NaOCl will be used
  Other Names: HEBP/NaOCl
  Arms: Etidronic acid/ Sodium Hypochlorite (HEBP/NaOCl)
Drug: Maleic acid — Final irrigation of root canal treatment procedure will be done with 5ml of maleic acid for 1min.
  Other Names: MA
  Arms: Maleic acid (MA)

SUMMARY:
The basic aim of root canal treatment is to reduce the microbial content and prevent further recontamination in the canal. Every tooth has a variable, complex canal anatomy consisting of ramifications, accessory and lateral canals. Instrumentation alone cannot reach all the areas for cleaning.The objectives of this research study is to observe and compare the effect of irrigation with smearOFF , etidronic acid/ hypochlorite and other irrigants on sealer penetration and dentin erosion of root dentin by using scanning electron microscope (SEM) and Energy Dispersive X-Ray Analysis (EDX).

Hundred extracted premolar teeth is subjected to root canal instrumentation. The endodontic procedure is done with protaper gold files. Initial irrigation is done by 5% sodium hypochlorite. Samples are divided into five groups. Each group consists of twenty single rooted premolars based on final irrigation regimen. There will be four experimental groups which are as follows (1) 17% EDTA (2) SmearOFF 3) Maleic acid (4) HEBP/NaOCL. Whereas, saline will be the control group. After the preparation and final irrigation of all teeth with experimental irrigants, sterile saline is used to flush all canals and dried using paper points. After final irrigation teeth are further divided into two groups (A) Sealer penetration (B) Dentin erosion. In both the groups standardization of root length, cleaning and shaping procedure are the same. For sealer penetration, obturation is done by warm vertical using AH plus sealer. Samples are incubated at 37º Celsius (°C) and 100% humidity for 7 days. The samples are marked and divided into three horizontal section at 2mm, 5mm and 8mm. Using SEM, measure the maximum depth of sealer penetration on each side that is buccal, lingual, mesial and distal and take the mean for each section of sample. For dentin erosion (B) samples are divided sagitally & buccolingually into two halves. The half containing the most visible part of apical area is taken and than examined using EDX. One-Way ANOVA-test will be used to compare mean values of multiple groups. Tukey's post hoc test will be used to determine the group with significance at P≤0.05. Two observers will evaluate the results using kappa statistics.

DETAILED DESCRIPTION:
Data Collection Extracted permanent premolars were collected from the department of Oral and maxillofacial surgery at Dow Dental College ( DDC,DUHS ) and Dr. Ishrat-ul-Ebad Khan Institute of Oral Health Sciences (DIKIOHS, DUHS). Following extraction, teeth were cleaned with tap water for all visible debris and stored in 0.1 % thymol at 4 C until further use.

METHODOLOGY

Extracted permanent premolars were collected from the department of Oral and maxillofacial surgery at Dow Dental College ( DDC,DUHS ) and Dr. Ishrat-ul-Ebad Khan Institute of Oral Health Sciences (DIKIOHS, DUHS). Teeth were cleaned with the help of ultrasonic scaler for any visible debris,soft tissue remnants and calculus and later examined under dental operating microscope for any visible crack or fracture. Teeth with presenting fracture, craze lines, developmental defects were discarded in accordance to the exclusion criteria. Digital periapical radiographs (PA) at three different angulations (45, 90 and 120) were taken to confirm the presence of a single straight canal within the root. After fulfilling the above mentioned criteria, hundred teeth were selected and stored in 0.1% thymol at 4C until further use.

Preparation of solutions:

1. Thymol = 1grams of thymol crystals were taken and dissolve it in 50ml ethanol. After dissolution, this solution was made upto 1 litre by distilled water.
2. 7 % Maleic acid = 7grams of maleic acid in powder form was dissolve in 100ml of distilled water to get 7% maleic acid.
3. 18 % Etidronic acid / 5.25 % sodium hypochlorite = For 18%, take 75 ml of standard solution and add 175 ml of distilled water in a volumetric to make total 250 ml HEBP. Both irrigants were mixed in 1:1 ratio. So, 250 ml of etidronic acid were mixed in 250 ml of sodium hypochlorite.

Sample Preparation All samples were prepared by a single operator using the following protocol. A standardized root length of 16mm was measured with the help of a Vernier caliper. After standardization the teeth were decoronated with diamond disc in slow speed hand piece . Access opening was performed using diamond round bur attached to high speed handpiece (D&G). The canal was explored using a 10 K-file (Mailefer/Dentsply) until its tip became visible at the apical foramen. Then, the working length was established as 1 mm shorter than the anatomical apical foramen. After that the apex was sealed by hot glue to simulate the in-vivo closed apex condition. Canal was prepared by using ProTaper gold (Dentsply-Sirona Switzerland). Standard sequence of files were used. Shaping files SX , S1 , S2 and finishing files F1 , F2 and F3 were used. A 30 guage side vented needle was used for irrigating 5.25 % NaOCl after every consecutive files. After cleaning and shaping with the above mentioned files, all teeth were divided into five groups.

Group Allocation The samples were randomly allocated into five groups. Four experimental and one control group. A computer-generated sheet (MS Excel) was used for randomization.

Group 1: Ethylene diamine tetra acetic acid (EDTA); (n = 20) Group 2 : SmearOFF; (n = 20) Group 3 : Maleic acid (MA); (n = 20) Group 4 : Etidronic acid / Hypochlorite (HEBP/ NaOCl); (n = 20) Group 5: Saline; (n=20)

In each group final irrigation protocol would be as follows

1. Group 1: EDTA = 5.25% NaOCl was used during instrumentation and 5ml of EDTA used for 1min as a final rinse.
2. Group 2: smearOFF = 5.25% NaOCl was during instrumentation and 5ml of smearOFF as a final rinse.
3. Group 3: Maleic acid = 5.25% NaOCl was during instrumentation and 5ml MA for 1 min as a final rinse was used
4. Group 4: Etidronic acid/ hypochlorite =1:1 mixture of 18 % HEBP / 5.25 % NaOCL was used during instrumentation and the same mixture as a final rinse for 1min

4. Group 5: Saline = 0.9 % solution was used during instrumentation and as a final rinse for 1min

The above mentioned experimental groups (Group 1: EDTA, Group 2: SmearOFF, Group 3: MA, Group 4: HEBP/NaOCl were rinsed with saline to create an isotonic environment. After final irrigation all the canals were dried with absorbent paper points. From here, all samples were divided into two groups: sealer penetration and dentin erosion.

Sample preparation for sealer penetration:

From each experimental and control group teeth were randomly selected and obturated using warm vertical condensation technique. After the canals had been dried obturation was performed using warm vertical condensation technique using AH plus sealer. The pre-fitted cone was lightly coated with AH plus sealer and placed into the canal; then, a heated plugger was activated and placed to a point 4-5 mm short of the working length and removed the coronal portion of master cone. Next, down-pack was performed. The remaining root canal was backfilled by using an injectable gutta-percha system (EQ-V) and vertical compaction was performed. Coronal part was sealed with Glass ionomer cement. Samples were kept at 37 °C and 100 % humidity for 7 days in an incubator to allow complete setting of the sealer. After 7 days the samples were taken out from incubator. The teeth were then embedded in epoxy resin moulds to form resin blocks of uniform dimensions.

Slides preparation After the resin was completely set, the samples were transversely sectioned at 2mm ( apical third ), 5 mm( middle third) and 8 mm (coronal third ) from the apex with the help of 0.3 mm blade used in diamond cutting saw ( Leco VC-50). Three sections with the thickness of 1mm each were obtained. Finishing was done by the help of silicone carbide sand paper and polishing was done using polishing machine. To remove the (in) organic debris, the specimens were cleaned in a bath with 15% EDTA for 2 minutes and then 3% NaOCl for 2 minutes. Samples were placed in sunlight for 24 hours inorder to have moisture free samples.

Analysis of sealer penetration into dentinal tubules

Sectioned teeth were marked at 2mm, 5mm and 8mm. Then specimens were mounted on metallic stubs and titanium-sputtered in Auto Fine Coater: JEC-3000FC. Coating was done on 20mA current for 30 seconds. Under scanning electron microscope (SEM JAPAN) model no JSM-IT 100 software:In touch scope, photomicrographs were taken. A blind independent observer examined samples for dentinal tubule penetration of sealers at three levels - 2,5 and 8 mm from the root apex. Of each sample one photomicrograph most representative of the section was taken from root-sealer interface at a magnification of 550x. On each of these photomicrographs, the minimum and maximum depth of sealer penetration in the tubules was measured.

Sample preparation for Dentin erosion

From each experimental groups 50 teeth were randomly selected. After performing cleaning and shaping, all the canals were dried with absorbent paper points. Two longitudinal grooves were prepared on the buccal and lingual surfaces of each root using a diamond disc without penetrating the canals. The roots were split into two halves using chisel and mallet. The half containing the most visible part of the canal was taken for evaluation. Then, the samples were marked at 2mm (apical third), 5mm (middle third) and 8 mm (coronal third) from the apex.

Analysis of Dentin erosion

Coating of the samples was done with platinum coater for evaluation under SEM. Then the samples were examined by SEM at x2000 magnification. Photomicrographs were taken at each third. Scoring of photomicrographs were done according to Torabinejad criteria by two independent observers. After that EDX analysis was done to determine total content of calcium and phophorus and the alteration in Ca/ P caused by various irrigants.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent single rooted premolars with single canal.
2. Sound teeth with mature apices.
3. Teeth extracted for orthodontic purpose.
4. Age between 17 -25 years (male or female)

Exclusion Criteria:

1. Intracanal calcification or pulp stones.
2. Root dilacerations and developmental defects. 3 Caries, fracture or cracked teeth.

4. Previously endodontically treated teeth or restorations. 5. Root resorption.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Sealer penetration | 4 months
  Samples were studied for dentinal tubule penetration by Scanning electron microscope (SEM) .They were evaluated at three levels coronal, middle and apical third by blinded independent observer. For each sample image, maximum linear depth of sealer penetration was measured in micrometers circumferentially at four locations (buccal, lingual, mesial and distal) . After recording four circumferential readings, final mean sealer penetration was calculated for each sample in micrometers
Dentin erosion | 2 months
  The erosion in the coronal, middle and apical third of the root canal walls were measured by scanning electron microscope (SEM). Photomicrogrpahs were scored by two independent investigators who were unaware of the groups using the scale suggested by Torabinejad et al score 1: No erosion, all tubules exhibited a normal appearance and size. Score 2: Moderate erosion, the peritubular dentin was eroded. Score 3: Severe erosion, the intertubular dentine was destroyed and the tubules were connected to each other.
  Chemical characterization (mass %) was performed by Energy Dispersive Xray spectroscopy (EDX).. All samples were then subjected to EDX analysis to determine total calcium (Ca) and phosphorus (P) content and the alteration in Ca/ P ratio on the root third of each group. The mineral content was not determined before the treatment of each sample because this analysis requires a destructive method. Thus, it is likely that the mineral content differed between all teeth

CONTACTS AND LOCATIONS:
Overall Officials: Sehrish Zubair, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan